CLINICAL TRIAL: NCT00752973
Title: Phase II, Multi-Center, Open-Label, Safety and Tolerance Study of a Novel Malathion Formulation in Infants and Toddlers With Pediculosis Capitis
Brief Title: Safety and Tolerability of a Novel Malathion Formulation in Children Age 6-24 Months With Head Lice
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MALG-0813
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-07

CONDITIONS: Pediculosis
Keywords: Head Lice
MeSH Terms: conditions — Lice Infestations | interventions — Malathion; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment arm (Experimental): MALG treatment
  Interventions: Drug: MALG (malathion) Treatment

INTERVENTIONS:
Drug: MALG (malathion) Treatment — MALG applied for 30 minutes
  Other Names: Novel malathion formulation

SUMMARY:
In a previous phase II study, the safety and efficacy of a novel formulation of malathion 0.5% was evaluated in patients 2 years of age and older. Based on the results of that study, this formulation is currently in a phase III study for that population.

The current study will use blood markers and clinical evaluations to determine the safety and tolerability of this formulation when used in children 6-24 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed active head lice infestation

Exclusion Criteria:

* Allergy to pediculicides or hair care products
* Scalp conditions other than head lice
* Previous head lice treatment within the past 4 weeks
* Current antibiotic treatment

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Investigator Site, Bentonville, Arkansas
  - Investigator Site, Jonesboro, Arkansas

REFERENCES:
- [Result] Meinking TL, Vicaria M, Eyerdam DH, Villar ME, Reyna S, Suarez G. A randomized, investigator-blinded, time-ranging study of the comparative efficacy of 0.5% malathion gel versus Ovide Lotion (0.5% malathion) or Nix Creme Rinse (1% permethrin) used as labeled, for the treatment of head lice. Pediatr Dermatol. 2007 Jul-Aug;24(4):405-11. doi: 10.1111/j.1525-1470.2007.00460.x. PMID 17845167

RESULTS

PARTICIPANT FLOW:
Groups:
- Malathion Gel 0.5% Treatment Arm: Malathion Gel 0.5% treatment
  MALG (Malathion Gel 0.5%) Treatment: MALG applied for 30 minutes
Period: Overall Study
Arm/Group | Malathion Gel 0.5% Treatment Arm
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- MALG Treatment Arm: MALG treatment
  MALG (malathion) Treatment: MALG applied for 30 minutes
Arm/Group | MALG Treatment Arm
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: months] | 17.5 (4.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 1
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Change in Cholinesterase Level at 1 Hour (Day 0).
Description: Each patient (aged 6 - 24 months) was assessed at 1 hour (Day 0). The mean percent change (reduction) in plasma and RBC cholinesterase activity from baseline to 1 hr after application was calculated and accompanied by 95% confidence intervals.
  If the half-widths of the derived confidence intervals are sufficiently narrow, it will demonstrate that any observed reductions in plasma and RBC cholinesterase activity fall within established safety guidelines.
  Concentration of RBC-cholinesterase (RBC-ChE) and plasma cholinesterase were obtained at baseline, at 1 hr (Day 0) and at 24 hrs (Day 1) after the application of the treatment.
  Mean percent change (reduction) = (Post treatment value - Baseline)/ Baseline x100.
Time Frame: Change from Baseline to 1 hour
Population: 10 subjects with obtained blood sample. subject 01-003: Study coordinator was unable to obtain blood sample post treatment at Visit 1, Day 0.
  subject 01-004: At Visit 1 Day 0 (post treatment), Blood sample could not be obtained even after two attempts.
Measure: Mean (95% Confidence Interval); unit: percentage change in cholinesterase
Groups:
- MALG (Malathion Gel, 0.5% )Treatment Arm: MALG (Malathion Gel, 0.5% ) treatment
  MALG (Malathion Gel, 0.5% ) Treatment: MALG applied for 30 minutes
  Two subjects had out of range RBC cholinesterase values. One subject had out of range (low) value at baseline and One subject had out of range (low) value 1 h post treatment. Both these values were considered to be not clinically significant by the investigator.
Arm/Group | MALG (Malathion Gel, 0.5% )Treatment Arm
Number analyzed (Participants) | 10
percentage change in cholinesterase
  Plasma | -1.8 [-3.9 to 0.4]
  RBC cholinesterase | -0.5 [-3.5 to 2.6]

2. Primary Outcome: Participants With a Change in Cholinesterase Level at 24 Hrs (1 Day).
Description: Each patient was assessed at Day 1 and the mean percent reduction in plasma and RBC cholinesterase activity from baseline to 24 hr after application was calculated and accompanied by 95% confidence intervals.
  Concentration of RBC-cholinesterase (RBC-ChE) and plasma cholinesterase were obtained at baseline, at 1 hr (Day 0) and at 24 hrs (Day 1) after the application of the treatment.
  Mean percent reduction = (Post treatment value - Baseline)/ Baseline x100.
Time Frame: Change from baseline to 24 hrs (1 day)
Population: 11 subjects with obtained blood sample. subject 01-004: At Visit 2, Day 1 Lab could not perform testing due to sample not suitable for testing. Because only 2ml blood was able to collected after multiple attempts.
Measure: Mean (95% Confidence Interval); unit: percentage change in cholinesterase
Groups:
- MALG (Malathion Gel, 0.5% )Treatment Arm: MALG (Malathion Gel, 0.5% ) treatment
  MALG (Malathion Gel, 0.5% ) Treatment: MALG applied for 30 minutes
  A subject had out of range (low) RBC cholinesterase value 1 h post treatment. This value was considered to be not clinically significant by the investigator.
Arm/Group | MALG (Malathion Gel, 0.5% )Treatment Arm
Number analyzed (Participants) | 11
percentage change in cholinesterase
  Plasma Cholinesterase | -1.7 [-5.0 to 1.7]
  RBC Cholinesterase | 1.4 [-1.8 to 4.6]

3. Primary Outcome: Participants With the Clinical Evidence of Cholinesterase Inhibition
Description: Participants with any of the following symptoms of cholinesterase inhibition as numbered below were considered to have Clinical evidence of cholinesterase inhibition.
  1. Abnormal heart rate.
  2. Diarrhea or abdominal cramps.
  3. Inappropriate sweating.
  4. Pupillary miosis (constriction).
  5. Respiratory difficulty such as chest tightness or wheezing.
  One participant had wheezing as medical history which continued without increase in severity throughout the treatment.
Time Frame: at Baseline
Measure: Number; unit: percentage of participants
Groups:
- MALG (Malathion Gel, 0.5% )Treatment Arm: MALG (Malathion Gel, 0.5% ) treatment
  MALG (Malathion Gel, 0.5% ) Treatment: MALG applied for 30 minutes
  Subjects who reported signs or symptoms of cholinesterase inhibition pre treatment
Arm/Group | MALG (Malathion Gel, 0.5% )Treatment Arm
Number analyzed (Participants) | 12
percentage of participants | 8.3

4. Primary Outcome: Participants With the Clinical Evidence of Cholinesterase Inhibition
Description: Participants with any of the following symptoms of cholinesterase inhibition as numbered below were considered to have Clinical evidence cholinesterase inhibition :
  1. Abnormal heart rate.
  2. Diarrhea or abdominal cramps.
  3. Inappropriate sweating.
  4. Pupillary miosis (constriction).
  5. Respiratory difficulty such as chest tightness or wheezing.
  One participants had wheezing as medical history which continued without increase in severity throughout the treatment.
Time Frame: at 1 hr (Day 0)
Measure: Number; unit: percentage of participants
Arm/Group | MALG (Malathion Gel, 0.5% )Treatment Arm
Number analyzed (Participants) | 12
percentage of participants | 8.3

5. Primary Outcome: Participants With the Clinical Evidence of Cholinesterase Inhibition
Description: Participants with any of the following symptoms of cholinesterase inhibition as numbered below were considered to have Clinical evidence of cholinesterase inhibition :
  1. Abnormal heart rate.
  2. Diarrhea or abdominal cramps.
  3. Inappropriate sweating.
  4. Pupillary miosis (constriction).
  5. Respiratory difficulty such as chest tightness or wheezing.
  One participants had wheezing as medical history which continued without increase in severity throughout the treatment.
Time Frame: at 24 hrs (Day 1)
Measure: Number; unit: percentage of participants
Arm/Group | MALG (Malathion Gel, 0.5% )Treatment Arm
Number analyzed (Participants) | 12
percentage of participants | 0

6. Primary Outcome: Participants Clinically Cured of Head Lice 14 Days After Last Treatment
Description: No live lice (including adults and nymphs) and nits at Day 7±1 and final lice assessment on either Day 14 (subjects not requiring retreatment) or Day 21 (for retreated subjects).
Time Frame: Day 7±1 and Day 14 or Day 21
Population: No statistical analysis provided for Clinical Cure
Measure: Number; unit: participants cured of lice
Arm/Group | MALG (Malathion Gel, 0.5% )Treatment Arm
Number analyzed (Participants) | 12
participants cured of lice | 12

7. Secondary Outcome: Evaluation of the Local Safety of Malathion Gel, 0.5% Based Upon Reported Adverse Events and Observed Scalp Reactions.
Description: To evaluate the safety of Malathion Gel, 0.5% based upon reported adverse events and observed scalp reactions. Additional safety assessments included eye Irritation.
Time Frame: Participants were followed for a minimum of 14 days (1 treatment) and a maximum of 21 days (2 treatments)
Population: A total of 12 subjects were enrolled. All of them used the study drug for at least one dose of the treatment. At Day 0 the study drug was to be used. At Day 7 if subject presented with live lice they were provided a second treatment. The subjects may used it for 1 (for subjects not requiring retreatment) or 2 (for retreated subjects).
Measure: Number; unit: participants
Arm/Group | MALG (Malathion Gel, 0.5% )Treatment Arm
Number analyzed (Participants) | 12
participants
  No sign of irritation | 11
  Slight noticeable erythema + slight infiltration | 1
  No conjunctival irritation | 12

ADVERSE EVENTS:
Time Frame: 22 months
Arm/Group | MALG Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MALG Treatment Arm (N=12)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No